CLINICAL TRIAL: NCT00098800
Title: A Multicenter Randomized Double-Blinded Trial for Chemoprevention of Ovarian Cancer: Modulation of Biomarkers and Spectral Properties Using Contrast Enhanced Ultrasound in High-Risk Women Using Fenretinide (4-HPR)
Brief Title: Fenretinide in Preventing Ovarian Cancer in Participants Who Are at High Risk for Developing Ovarian Cancer and Planning to Undergo Surgery to Remove the Ovaries
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Arizona (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Allocation: Randomized | Masking: Double | Purpose: Prevention
Other Study IDs: CDR0000396796; P30CA016672 (NIH); UARIZ-GYN-01021; UARIZ-HSC-02190; MDA-GYN-01021
Record Dates: First submitted 2004-12-08; First posted 2004-12-09 (Estimated); Last update posted 2010-03-24 (Estimated); Status verified 2006-11

CONDITIONS: brca1 Mutation Carrier; brca2 Mutation Carrier; Ovarian Cancer
Keywords: ovarian epithelial cancer; BRCA1 mutation carrier; BRCA2 mutation carrier
MeSH Terms: conditions — Ovarian Neoplasms; Carcinoma, Ovarian Epithelial | interventions — Fenretinide

INTERVENTIONS:
Drug: fenretinide

SUMMARY:
RATIONALE: Chemoprevention is the use of certain drugs to keep cancer from forming, growing, or coming back. The use of fenretinide may prevent ovarian cancer.

PURPOSE: This randomized clinical trial is studying how well fenretinide works in preventing ovarian cancer in participants who are at high risk of developing ovarian cancer and planning to undergo surgery to remove the ovaries.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Compare the induction of apoptosis (as determined by TUNEL) in the ovarian epithelial and stromal cells of participants at high risk for ovarian cancer treated with fenretinide vs placebo.

Secondary

* Compare modulation of several intermediate markers (TGFβ, BAX, Ki-67, ER, PR, RARβ, TGFβRI, TGFβRII, p21, p53, FAS, and FASL) in participants treated with these regimens.
* Compare early microvascular changes, using contrast-enhanced ultrasound, in participants treated with these drugs.
* Determine whether the use of contrast agents could indicate changes in ovarian size and architecture that may be assessed as potential surrogates for preventive effect in these participants.
* Determine the feasibility of future chemoprevention trials for ovarian cancer.
* Determine the toxicity of fenretinide in these participants.
* Compare the microvascularity index and ovarian volume of participants treated with these drugs.
* Correlate areas of increased microvascularity and other abnormalities with pathology findings obtained at oophorectomy in participants treated with these drugs.

OUTLINE: This is a randomized, double-blind, placebo-controlled, multicenter study. Participants are randomized to 1 of 2 treatment arms.

* Arm I: Participants receive oral fenretinide once daily.
* Arm II: Participants receive oral placebo once daily. In both arms, treatment continues for 6-8 weeks in the absence of unacceptable toxicity.

Within 5 days after completion of fenretinide or placebo, participants undergo bilateral salpingo-oophorectomy.

Participants are followed at 6 weeks.

PROJECTED ACCRUAL: A total of 40 participants (20 per treatment arm) will be accrued for this study within 4 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* At high risk for developing ovarian cancer, meeting 1 of the following criteria:

  * Family history of ovarian cancer, defined as ≥ 1 first-degree relative diagnosed with ovarian cancer before 50 years of age
  * Family history of ovarian cancer, defined as ≥ 1 first-degree relative diagnosed with ovarian cancer at any age AND ≥ 1 first- or second-degree relative diagnosed with breast or ovarian cancer at any age
  * Positive BRCA1/BRCA2 test
* Planning to undergo prophylactic bilateral oophorectomy

PATIENT CHARACTERISTICS:

Age

* 30 and over

Performance status

* Zubrod 0-1

Life expectancy

* At least 12 months

Hematopoietic

* Not specified

Hepatic

* Bilirubin ≤ 1.5 times upper limit of normal (ULN)
* SGOT ≤ 1.5 times ULN
* Alkaline phosphatase ≤ 1.5 times ULN
* No history of liver disease*
* No cholestatic jaundice
* No hepatic adenomas NOTE: *For patients undergoing contrast enhanced ultrasound

Renal

* BUN normal
* Creatinine normal

Cardiovascular

* No history of a congenital heart defect creating a bi-directional or right-to-left shunt*
* No history of congestive heart failure*
* No thrombophlebitis
* No thromboembolic disease
* No cerebral vascular disease
* No coronary artery disease NOTE: *For patients undergoing contrast enhanced ultrasound

Pulmonary

* No history of pulmonary hypertension*
* No history of pulmonary emboli*
* No history of severe emphysema* NOTE: *For patients undergoing contrast enhanced ultrasound

Other

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective barrier contraception
* Thyroid stimulating hormone normal
* T4 normal
* Triglycerides ≤ 1.5 times ULN
* No malignancy within the past 5 years except breast cancer or basal cell or squamous cell skin cancer

  * No evidence of recurrent disease
* No known or suspected hypersensitivity to blood, blood products, or albumin
* No undiagnosed genital bleeding
* No history of pancreatitis
* No uncontrolled diabetes
* No other severe underlying chronic disease
* No concurrent alcohol use (> 3 drinks/day or equivalent)

PRIOR CONCURRENT THERAPY:

Biologic therapy

* Not specified

Chemotherapy

* At least 3 months since prior chemotherapy for breast cancer

Endocrine therapy

* No concurrent selective estrogen-receptor modulators, including raloxifene
* No concurrent aromatase inhibitors

Radiotherapy

* Not specified

Surgery

* See Disease Characteristics

Other

* More than 3 months since prior therapeutic oral or topical vitamin A derivatives (e.g., isotretinoin)
* No other concurrent investigational agents
* No concurrent cyclooxygenase-2 (COX-2) inhibitors
* No concurrent oral vitamin A or ascorbic acid (vitamin C) supplements > recommended daily requirement (10,000 IU for vitamin A and 75 mg for vitamin C)

Min Age: 30 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2004-10; Primary Completion 2006-08 (Actual); Study Completion 2006-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Molly A. Brewer, MD, DVM, MS, Principal Investigator — University of Arizona
Locations (1):
- Arizona Cancer Center at University of Arizona Health Sciences Center, Tucson, Arizona, United States